CLINICAL TRIAL: NCT01178762
Title: The Effect of Oral Azithromycin in the Treatment of Chlamydial Conjunctivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yan-Ming Chen / Yu-Chih Hou, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200709013R
Record Dates: First submitted 2008-08-31; First posted 2010-08-10 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-09

CONDITIONS: Chlamydial Conjunctivitis
Keywords: Oral Azithromycin; Chlamydial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Inclusion | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Observation (Experimental)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Oral Azithromycin in the Treatment of Chlamydial Conjunctivitis
  Other Names: zithromax(Pfizer)

SUMMARY:
Chlamydia trachomatis is one of the major causes of sexually transmitted disease and also the leading infectious cause of blindness in the world.Treatment of C. trachomatis eye infection has involved for a long time. The efficacy of single dose azithromycin has already been demonstrated as effective in the treatment of both trachoma and adult inclusion conjunctivitis.However, in our clinical experience, some patients of chlamydial conjunctivitis may require augmented single dose azithromycin treatments before C. trachomatis is eradicated. In this way, we would like to known the efficacy of single dose and augmented single dose azithromycin in the treatment of chlamydial conjunctivitis.

DETAILED DESCRIPTION:
Medical records of patients with clinically suspected chlamydial conjunctivitis between January 1, 2006 and December 31, 2006 at one cornea specialist's (Y.C.H) out-patient clinic were retrospectively reviewed. At this clinic, patients of both sexes with acute, chronic or recurrent follicular conjunctivitis with the symptoms and signs of chlamydial conjunctivitis suspected were tested for Chlamydia direct fluorescent antibody (DFA) tests and arranged for next time out-patient clinic follow up 1-2 weeks later. The patients who attended the follow up visit with positive DFA results were treated with oral azithromycin. These patients received a single dose oral azithromycin (400mg~1000mg, according to their age and body weight) once a week for consecutive two weeks. Repeated DFA examinations were performed 4 to 6 weeks later. If the DFA examinations still showed positive results, augmented single dose oral azithromycin once a week for one week was given again till the DFA showed negative results. The occurrence and frequency of adverse events recorded in the medical charts were reviewed as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients of clinically chlamydial conjunctivitis suspected and proven by direct fluorescent antibody(DFA)results

Exclusion Criteria:

* Patients with pregnancy or lactation, history of allergy to macrolides, evidence or history of hepatic, renal, hematological or cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chih Hou, MD, Study Director — National Taiwan University Hospital; Fung-Rong Hu, MD, Study Director — National Taiwan University Hospital; Yan-Ming Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Publication provided — http://www.ncbi.nlm.nih.gov/pubmed/19893589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with clinically suspected chlamydial conjunctivitis at the outpatient clinic of Dr Hou at National Taiwan University Hospital (NTUH) between 1 January 2006 and 31 December 2006 were included
Pre-assignment Details: Patients with symptoms and signs of chlamydial conjunctivitis suspected were tested for Chlamydia direct fluorescent antibody tests. The patients with positive results were treated with oral azithromycin,except those who were pregnant, lactating,with a history of allergy to macrolides or hepatic, renal,hematological or cardiovascular disease .
Groups:
- Azithromycin: DFA positive chlamydial conjunctivitis patients were orally administered azithromycin (400mg~1000mg, according to their age and body weight) once a week for consecutive two weeks, and the DFA tests were repeated 4 weeks after the treatment. If the DFA tests still showed positive results, an additional dose of azithromycin was orally administered, and another DFA test was performed again 4 weeks later. The augmented treatment with oral azithromycin (administration of one oral dose followed by DFA testing 4 weeks later) was continued until the DFA tests showed negative results.
Period: Overall Study
Arm/Group | Azithromycin
Started | 42
Completed | 27
Not Completed | 15
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 28
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Region of Enrollment [Number; unit: participants]
  Taiwan | 42

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With Negative Chlamydia Direct Fluorescent Antibody (DFA) Test Results After Oral Azithromycin Treatments
Description: We performed direct fluorescent antibody (DFA) tests for Chlamydia by swabbing across the lower and upper tarsal conjunctiva four times after topical application of 0.5% proparacaine. All of the DFA tests were examined by the same experienced microbiologist who was masked to the identities and clinical conditions of the patients. Each DFA slide was read under a fluorescent microscope and was observed for discrete fluorescent chlamydial elementary bodies (EBs).The DFA test was considered positive if above 10 EBs were counted per high-power field.
Time Frame: 4 weeks, 8 weeks and 12 weeks after the first dose of the medication
Population: Only participants with confirmed DFA tests are counted in the results below. Participants with confirmed negative DFA tests subsequently stopped treatment and were not retested. Participants lost to follow-up are counted as not having a confirmed DFA negative test
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 42
participants | 27

ADVERSE EVENTS:
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No